CLINICAL TRIAL: NCT03891095
Title: Oxytocin and Dopamine's Effect on Vicarious Optimism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, ma, yina, Principal Investigator, Beijing Normal University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OT-DA-Vicarious optimism
Record Dates: First submitted 2019-03-17; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Oxytocin Group; L-DOPA Group; Placebo Group
Keywords: intranasal oxytocin; L-DOPA; Vicarious optimism
MeSH Terms: interventions — Oxytocin; Levodopa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intranasal oxytocin (Experimental): Oxytocin (OXT), a neuropeptide produced in the hypothalamus, is a key modulator of complex socioaffective responses including affiliation, social approach and attachment, stress and anxiety. Subjects receiving an intranasal spray of OXT (24 IU or 40.32 mg; Syntocinon-spray; Novartis, Switzerland)
  Interventions: Drug: Oxytocin; Drug: Placebos
- L-DOPA (Experimental): L-DOPA, a neuropeptide who is a key modulator of complex socioaffective responses including reward, social decision making, learning. Subjects receiving 187.5 mg Madopar (L-DOPA treatment, including 150 mg L-3,4-dihydroxyphenylalanine, together with 37.5 mg benserazide, which promotes higher levels of dopamine in the brain while minimizing side effects from peripheral dopamine)
  Interventions: Drug: L-DOPA; Drug: Placebos
- Placebo (Placebo Comparator): Participants in the Placebo group received spray and oral placebos. 24 IU saline (spray placebo) 187.5 mg calcium carbonate (oral placebo)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Oxytocin — intranasally administrated
  Arms: Intranasal oxytocin
Drug: L-DOPA — orally administered
  Arms: L-DOPA
Drug: Placebos — intranasally administrated and orally administered

SUMMARY:
To investigate the effect of intranasal Oxytocin and L-DOPA's effect on vicarious optimism.

DETAILED DESCRIPTION:
The current study adopted a double-blind, double-dummy, placebo-controlled mixed design, with Treatment (oxytocin, dopamine, and placebo) as a between-subjects factor, and Target (self, friend, and an identifiable stranger) and Feedback (desirable vs. undesirable) as within-subjects factors. Upon arrival, participants first completed a set of questionnaires, including mood measurements and other questionnaires related to optimistic or prosocial tendency. Participants then self-administered with the pharmacological challenge 40 min before the main task, i.e., the belief updating task where participants indicated and updated their beliefs about the future of oneself, a gender-matched best friend, and a gender-matched identifiable stranger. At the end, participants completed the mood measurement again, as well the debriefing questionnaires which designed to measure their beliefs about the experimental process.

For the vicarious optimism task, participants completed three blocks of the two-session belief updating task where they were asked to estimate the likelihood of adverse life events happening to three targets: themselves (referred as Self), a gender-matched best friend (referred as Friend), and an identifiable stranger (whose name, brief description and picture were presented to the participants to get familiar with before the estimation, such as "The stranger is Zhexing, a 25-year-old male, Chinese"; referred as Stranger).

Participants completed two estimation sessions for one target before beginning with the next target, and the order of targets was counterbalanced across participants within each group. For the first session of each target block, participants were first presented with 30 different adverse life events (in a random order) and estimated the likelihood of each event happening to the target in the future (the 1st estimation, referred to as E1) on a self-paced basis. Participants were then presented with the probability of each event occurring to an average person in a similar environment (Feedback) for 2s. In the second session, participants estimated the likelihood of the same 30 events (in a random order) happening to the target person again without receiving feedback (the 2nd estimation, referred to as E2).

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* subjects with past or current psychiatric or neurological disorders

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — we opted to recruit only males for the present study.
Enrollment: 156 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Belief update value for self, friend and stranger | 40~70 minutes after drug administration
  In the vicarious optimistic bias task, participants would make first estimation about the happening likelihood for each event for themselves, friend, and stranger and then receive feedback about the general likelihood of each event happened in future. After all events first estimation, participants would estimate all the event again. So, for the belief update, we used the second estimation value to minus the first estimation value to get the update value, as well as calculating the update value in desirable condition (first estimation < feedback) and undesirable condition (first estimation < feedback). Then investigated the general belief updating (gBU) and optimistic belief updating (using desirableBU-undesirableBU) for the three target (self vs. friend vs. stranger) in three treatment groups (Oxytocin vs. L-DOPA vs. Placebo)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Normal University, Beijing, Beijing Municipality, China